CLINICAL TRIAL: NCT07156136
Title: A Phase 1 First-in-Human Study of the Safety and Efficacy of IMC-P115C as a Single Agent and in Combination With Standard of Care Agents in HLA-A*02:01 Positive Participants With Advanced PRAME Positive Cancers
Brief Title: Study of IMC-P115C in Advanced PRAME-Positive Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Immunocore Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMC-P115C-1005; 2023-509767-25 (Other: EU CTR)
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: PRAME Positive; Cancer; HLA-A*02:01-positive
Keywords: PRAME
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will include sequential assignment for non-randomized and randomized arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm A: IMC-P115C Monotherapy (Experimental): Participants receive IMC-P115C intravenous (IV) infusion
  Interventions: Drug: IMC-P115C

INTERVENTIONS:
Drug: IMC-P115C — IV infusion

SUMMARY:
Phase 1 First-in-human study of the safety and efficacy of IMC-P115C as a single agent and in combination with standard of care (SOC) agents in participants with advanced PRAME positive cancers. IMC-P115C is a half-life extended (HLE) ImmTAC targeting PRAME.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* HLA-A*02:01-positive
* Meeting PRAME-positive tumor testing requirements
* Metastatic or unresectable solid tumors
* Have received (or be receiving), relapsed from, be refractory to or intolerant of all therapies
* Male and female participants of childbearing potential who are sexually active with a non-sterilized partner must agree to use highly effective methods of birth control

Exclusion Criteria:

* Symptomatic or untreated central nervous system metastasis
* Bowel obstruction, perforation, or fistula formation within 3 months prior to the planned first dose of study treatment
* Ongoing ascites or effusion requiring recent drainages
* Significant ongoing toxicity from prior anticancer treatment
* Out-of-range laboratory values
* Clinically significant lung, heart, or autoimmune disease
* Ongoing requirement for immunosuppressive treatment
* Significant secondary malignancy
* Hypersensitivity to study drug or excipients
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with dose-limiting toxicities (DLT) | Up to ~16 months
Percentage of participants with adverse events (AE) | Up to ~16 months
Percentage of participants with serious adverse events (SAE) | Up to ~16 months
Percentage of participants with a dose interruption, reduction, or discontinuation | Up to ~16 months
  Percentage of participants with dosing changes or discontinuations.

SECONDARY OUTCOMES:
Best Overall Response (BOR) as determined by RECIST v1.1 per the Investigator. | Up to ~19 months
Duration of Response (DOR) as determined by RECIST v1.1 per the Investigator. | Up to ~19 months
Progression Free Survival (PFS) as determined by RECIST v1.1 per the Investigator. | Up to ~19 months
Overall Survival (OS) | Up to ~19 months
  OS is the time from first dose of study therapy until death due to any cause.
Change from baseline in lymphocyte counts | Up to ~19 months
  Change from baseline in lymphocyte counts
Changes in serum cytokine concentrations | Up to ~19 months
  Change from baseline in serum cytokine concentrations
IMC-P115C Plasma Concentration | Up to ~19 months
  IMC-P115C plasma concentration
Percentage of participants with anti-IMC-P115C antibody formation | Up to ~19 months

CONTACTS AND LOCATIONS:
Locations (13):
- Australia (3):
  - Cancer Research South Australia (CRSA), Adelaide
  - Linear Clinical Research ltd., Nedlands
  - Melanoma Institute Australia, Wollstonecraft
- France (3):
  - UNICANCER - Centre Leon-Berard (CLB), Lyon
  - Centre Hospitalier Universitaire (CHU) de Toulouse-Institut Universitaire du Cancer de Toulouse-Oncopole (IUCT-Oncopole), Toulouse
  - Institut Gustave Roussy, Villejuif
- Italy (3):
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione "G. Pascale", Napoli
- Spain (4):
  - Hospital Universitari Vall d Hebron, Barcelona
  - Institut Catala d'Oncologia (ICO) - Hospital Duran i Reynals, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - START Madrid - Hospital Universitario Fundación Jiménez Díaz, Madrid